CLINICAL TRIAL: NCT06188416
Title: Changes in Dynamic q Angle in Patients With Chronic Ankle Instability
Acronym: Dynamic knee v
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abdelmoniem Mohamed, Demonstrator, Cairo University
Other Study IDs: P.T.REC/012/004802
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Ankle Sprain Strain
Keywords: Kinetic chain; Ankle instability; Q-angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with CAI: Cases that reported previous experience of chronic ankle instability
- Cases without CAI: Cases that did not report any previous experience of chronic ankle instability

SUMMARY:
This study investigates the difference in dynamic Q-angle of patients with chronic ankle instability and those without.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged between 18 and 30 years.
* Subjects with a history of LAS for at least one year before the study onset, that required at least 1-day weight-bearing restriction.
* Subjects with a self-reported tendency of ≥2 giving way episodes during 6 months before enrollment in the study.
* Subjects with a perception that the injured ankle was chronically weaker, more painful, and/or less functional than the contralateral ankle before the first LAS.
* Subjects who scored less than 24 in the Cumberland Ankle Instability Tool (CAIT), a validated ankle instability specific questionnaire of 9 items, to determine if functional ankle instability is present.

Exclusion criteria

* Subjects who had bilateral LAS
* Subjects with a history of lower extremity injury, fracture, or surgery
* Subjects who participated in supervised or unsupervised ankle rehabilitation within a year before enrollment in the study
* Subjects with LAS within 3 months before participation
* Subjects with a history of knee pain during the last 6 months.
* Subjects diagnosed with knee osteoarthritis.

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: The participants from both genders aged between 18 and 30 years will be divided into 2 groups: a study group and a control group. The study group consists of 52 participants with chronic ankle instability, and the control group consists of 52 participants without chronic ankle instability, normal participants with no musculoskeletal disorders or history of knee disease and no obvious limb length discrepancy.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2023-11-26 (Actual); Study Completion 2023-12-03 (Actual)

PRIMARY OUTCOMES:
Dynamic Q-angle | 6 months
  Using dynamic knee valgus through the measurement of frontal plane projection angle

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Dokki, Giza Governorate, Egypt